CLINICAL TRIAL: NCT02222636
Title: The Clinical Research of Intranasal Dexmedetomidine Used in Plastic Surgery of Children : A Single Center ,Randomized ,Double-blinded, Controlled Study.
Brief Title: The Clinical Research of Intranasal Dexmedetomidine Used in Plastic Surgery of Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, wangqiang, department of anesthesijology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sedation wei
Record Dates: First submitted 2014-08-14; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: The Efficacy and Safety of Intranasal Dexmedetomidine
Keywords: The efficacy and safety of intranasal dexmedetomidine
MeSH Terms: interventions — Sevoflurane; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1,Normal saline,1 milliliter (Placebo Comparator): Patients will be assigned to receive intranasal normal saline 1 milliliter
  Interventions: Drug: Normal saline,1 milliliter; Drug: Anesthesia induction, 8% sevoflurane; Drug: Anesthesia maintenance, 2%~3% sevoflurane,fentanyl
- Group 2,dexmedetomidine 1μg.kg-1,1 milliliter (Experimental): Patients will be assigned to receive intranasal dexmedetomidine( 1μg.kg-1) 1 milliliter
  Interventions: Drug: Dexmedetomidine 1 μg.kg-1,1 milliliter; Drug: Anesthesia induction, 8% sevoflurane; Drug: Anesthesia maintenance, 2%~3% sevoflurane,fentanyl
- Group 3,dexmedetomidine 2μg.kg-1,1 milliliter (Experimental): Patients will be assigned to receive intranasal dexmedetomidine( 2μg.kg-1 )1 milliliter
  Interventions: Drug: Dexmedetomidine 2μg.kg-1,1 milliliter; Drug: Anesthesia induction, 8% sevoflurane; Drug: Anesthesia maintenance, 2%~3% sevoflurane,fentanyl

INTERVENTIONS:
Drug: Normal saline,1 milliliter — Normal saline,1 milliliter, 20 minutes before anaesthetic induction
  Arms: Group 1,Normal saline,1 milliliter
Drug: Dexmedetomidine 1 μg.kg-1,1 milliliter — Dexmedetomidine 1 μg.kg-1,1 milliliter,20 minutes before anesthesia induction
  Arms: Group 2,dexmedetomidine 1μg.kg-1,1 milliliter
Drug: Dexmedetomidine 2μg.kg-1,1 milliliter — Dexmedetomidine 2μg.kg-1,1 milliliter,20 minutes before anesthesia induction
  Arms: Group 3,dexmedetomidine 2μg.kg-1,1 milliliter
Drug: Anesthesia induction, 8% sevoflurane — Inhalation induction with 8% sevoflurane
Drug: Anesthesia maintenance, 2%~3% sevoflurane,fentanyl — 2%~3% sevoflurane,inhalation. fentanyl,2μg.kg-1.min-1,intravenous infusion

SUMMARY:
The purpose of this study is to explore the optimal protocol for dexmedetomidine used in children during perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Elective cleft lip and cleft palate repair surgery
* American Society of Anesthesiologists class I
* Aged between 6 months and 7 years old

Exclusion Criteria:

* Suspected or confirmed difficult airway
* History of upper respiratory tract infection with 1 month
* Combined with congenital heart disease
* Allergic to investigational products or with other contraindication
* Growth retardation or dysgnosia
* Central nervous system disease
* Serious infection
* Serious heart,brain,liver,kidney, pulmonary, and endocrine disease

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Sedation-Agitation Scale | The moment of entering operating room,20 minutes before anesthesia induction,10 minutes before anesthesia inducion,the moment of anesthesia induction
The pediatric anesthesia emergence delirium scale | The moment of entering operating room,and from discontinuation of inhalational anesthetics to the moment of patient's consciousness recovery,an expected average of 1 hour
Anesthesia induction time | From beginning of inhalating anesthetics to the moment of intubation
Anesthesia maintenance time | From the moment of intubation to the discontinuation of inhalational anesthestics
Recovery time | From discontinuation of inhalational anesthestics to the moment of patient's consciousness recovery, an expected average of 1 hour
Change from baseline in blood pressure during anesthesia | The moment of entering operating room,20 minutes before anesthesia induction,10 minutes before anesthesia inducion,the moment of anesthesia induction
Change from baseline in heart rate during anesthesia | The moment of entering operating room,20 minutes before anesthesia induction,10 minutes before anesthesia inducion,the moment of anesthesia induction
Change from baseline in respiratory rate during anesthesia | The moment of entering operating room,20 minutes before anesthesia induction,10 minutes before anesthesia inducion,the moment of anesthesia induction

SECONDARY OUTCOMES:
The alveolar concentration of inhalational anesthetics | the moment of anesthesia induction,the moment of intubation,before cutting skin